CLINICAL TRIAL: NCT05233137
Title: Enhancing Muscle Function After Exacerbations of COPD to Limit Its Impact on Physical Activity Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Prof. Dr, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S65813
Record Dates: First submitted 2022-01-11; First posted 2022-02-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1:1 allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PA coaching and exercise training (Experimental): Patients in this group will receive physical activity telecoaching as well as an exercise training program provided by a physiotherapist in primary care
  Interventions: Behavioral: PA coaching; Other: Exercise training
- PA coaching (Active Comparator): Patients in this group will receive physical activity telecoaching
  Interventions: Behavioral: PA coaching

INTERVENTIONS:
Behavioral: PA coaching — PA coaching: Patients receive a step counter together with a coaching application (m-PAC, AppsOnly, KU Leuven) installed on a smartphone. The step counter and coaching application are connected via Bluetooth. The coaching application has the goal of PA promotion as well as detecting any new AECOPD.
Other: Exercise training — Each session will include at least the following components:
  * Resistance training of the lower limbs: Exercises for 6 muscle groups using minimal (e.g. ankle weights or elastic resistance bands) or no (body weight) equipment are foreseen. Each exercise will be performed in 3 series of 8 repetitions.
  * Functional training: Sit to stand exercise and stair climbing. During the first 2 weeks of the exercise training program, at least 3 strength exercises and 1 functional exercise will be performed each session.
  Starting from the 3rd week of the exercise training program, whole body exercise training (interval training for walking, cycling, stair climbing and high knees) will be added. From this moment on, at least 1-2 whole body exercises and 2-3 strength and functional exercises will be performed during each physiotherapy session. By doing this, each session will consist of a minimum of 4 exercises in total.
  Arms: PA coaching and exercise training

SUMMARY:
Patients with COPD lose muscle strength during acute exacerbations of COPD (AECOPD) which interferes improving the recovery of physical activity (PA) after an AECOPD. Resistance training can reverse this process. An exercise training program with the focus on resistance training is essential in minimizing the long-term effects of AECOPD as it may help to accelerate the gain in PA in the weeks after an acute event. Therefore, it is important that such programs are embedded at the right moment (i.e. immediately after an AECOPD) and in a setting accessible to the patient (i.e. primary care). The efficacy and effectiveness of implementing such training programs will be assessed in the present study.

DETAILED DESCRIPTION:
The present study aims to:

1. Investigate whether an 8 week exercise training program provided in primary or community care enhances lower limb muscle strength in patients following an AECOPD;
2. Investigate whether such programs assist patients after an AECOPD to re-engage with a coaching intervention geared to long-term PA maintenance or improvement.

The secondary aim is to investigate how (repeated) AECOPD contribute to structural alterations in the skeletal muscle and how an exercise training program and PA can influence the deterioration in muscle fiber morphology and signals related to muscle atrophy.

Patients that experience a moderate or severe AECOPD will be recruited in the present multicentre randomised controlled trial (RCT).

Patients in this study will have at least 3 clinical visits:

* Post AECOPD treatment: screening and randomisation visit (V1)
* 8 weeks after randomisation (V2a and V2b*)
* 52 weeks after randomisation (V3a and V3b*)

  * If patients agree to have a muscle biopsy taken, a V2b and V3b will be added, so this does not interfere with other measurements. These visits will take place 1-2 weeks after V2a and V3a, respectively.

After the screening and randomisation visit (V1), the patient will be randomised in either the intervention group (PA coaching and exercise training) or the control group (PA coaching).

Patients in the intervention group will receive a first physiotherapy session during this first visit provided by the trained researchers (with a degree in physiotherapy) to get acquainted with the exercises. Information about the PA coaching will be given to all the patients. The intervention will be started after this visit and is provided by a physiotherapist in primary or community care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Smoking history (> or = 10 pack years)
* Experiencing a moderate (i.e. treated with short acting bronchodilatators plus antibiotics and/or oral corticosteroids or emergency room visit and reported impact on activities of daily living) exacerbation

Exclusion Criteria:

* More than 21 days after stopping the treatment for the AECOPD
* Presence of orthopaedic problems or other contra-indications not allowing to perform PA
* Participation in or planned to start a multidisciplinary pulmonary rehabilitation program
* Already participating in an intensive training program in the first 12 weeks in primary care with the aim of enhancing physical performance (maintenance programs are allowed)
* Unable to learn to work with a smartphone and Fitbit, as judged by the investigator
* Underwent major lung surgery (e.g. lung transplantation) or active on the lung transplantation list
* Lung volume reduction within 6 months before inclusion
* Having the current diagnosis of lung cancer or receiving active treatment for oncology

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Daily number of steps at 52 weeks | 52 weeks
  Change in daily mean step count 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Isometric quadriceps force | 8 weeks
  Isometric quadriceps strength of the right leg will be measured using the strain gauge device (Sauter Controls NV, Zellik, Belgium) with the hip and knee in 90° flexion. Four repetitions will be performed using standardized encouragement with the first attempt not being maximal and not counting as a possible best result. The best of the last three measurements will be used.

SECONDARY OUTCOMES:
Functional exercise capacity | 8 and 52 weeks
  Change in six-minutes walk distance between baseline and 52 weeks post randomization in the intervention group as compared to the control group. The six-minutes walk test will be performed with standardized encouragement to assess patients' functional exercise capacity. The best of two measurements will be used.
Isometric quadriceps force | 52 weeks
  Isometric quadriceps strength of the right leg will be measured using the strain gauge device (Sauter Controls NV, Zellik, Belgium) with the hip and knee in 90° flexion. Four repetitions will be performed using standardized encouragement with the first attempt not being maximal and not counting as a possible best result. The best of the last three measurements will be used.
Functional performance | 8 weeks and 52 weeks
  This will be evaluated using the SPPB. This test assesses lower extremity function and mobility. It consists of 3 subtests that are scored and points are added up:
  * 4-meter gait speed: To evaluate the patient's functional gait speed. The test is repeated twice. The best time of the 2 attempts is used for the rating. Cut-off: <0.3 m/s or ≥0.3 m/s.
  * 5 times sit to stand: This test quantifies the functional lower extremity strength. In this test, patients are asked to complete 5 cycles sit-to-stand as fast as possible from a 45 cm height chair. The participant may practice 1 repetition prior commencing the test. The time needed to perform 5 repetitions is noted. Cut-offs: ≤11.19 seconds (4 points); A higher score indicates a better functional performance.
Health related quality of life | 8 weeks and 52 weeks
  Change in health related quality of life wil be measured by the Chronic Respiratory Disease Questionnaire (CRDQ-SAS) (dyspnea domain):
  This disease specific questionnaire measures both physical and emotional aspects of the chronic respiratory disease. The questionnaire contains 20 items, spread over 4 domains (dyspnea, fatigue, emotional function and mastery). The MCID is reflected by a change in score of 0.5 on a 7-point scale for each of the CRDQ domains (28). Only the dyspnea domain will be used for this study. The self-administered standardized (CRDQ-SAS) version will be used. A higher score indicates a higher health related quality of life.
Health status | 8 weeks and 52 weeks
  Change in health status will be measured using the COPD Assessment Test (CAT):
  This validated 8-item questionnaire assesses the impact of the disease on a patient's health status. Scores range from 0 (good health status) to 40 (worse health status). The minimal clinical important difference (MCID) is a change of 2 points (19).
Patient experience of PA | 8 weeks and 52 weeks
  Change in patient experience of physical activity will be measured using the Patient Reported Outcome (PRO) -active (C-PPAC) questionnaire: a simple, valid and reliable 12-item questionnaire assessing PA from a patient's perspective reflecting on the past 7 days. The questionnaire investigates the experienced amount of and difficulty of PA as perceived by the patient. The 2 domain scores as well as the total score will be retrieved as outcomes. The clinical visit version will be used. A paper version of the questionnaire will be given along with the monitor. Subscores and total score are from 0 to 100, with higher score meaning less problems with daily life activities as reported by the patient
Change in high-density lipoprotein (HDL) | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Change in low-density lipoprotein (LDL) | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Change in total cholesterol | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Change in triglycerides | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient and triglycerides) and blood pressure
Change in blood pressure | 8 weeks and 52 weeks
  By taking the systolic and diastolic blood pressure of the patient at rest
Change in weight | 8 weeks and 52 weeks
  By taking the weight of the patient
Change in waist and hip circumference | 8 weeks and 52 weeks
  The waist and hip circumference will be measured and risk factors fasting blood sample (glucose level, insulin Hba1c)
Change in insulin | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Change in glucose level | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Change in Hba1c | 8 weeks and 52 weeks
  By taking a fasting blood sample of the patient
Day to day Physical Activity | 52 weeks
  Change in day to day data of PA will be assessed by a wearable. The patient receives a step counter (Fitbit) that can be worn on the wrist. The device provides direct feedback, expressed as the number of steps taken per day. The patient is asked to wear the step counter every day during the intervention and is invited to frequently verify the number of steps per day against the agreed goals.
Number of AECOPD | 52 weeks
  Number of AECOPD following the index AECOPD
Change in fiber type proportion of the m. vastus lateralis of the quadriceps muscle | 8 weeks (+1-2 weeks) and 52 weeks (+1-2 weeks)
  By analysing muscle microbiopsies of the quadriceps muscle immunostaining of the myosin heavy chain, only for patients giving their specific consent.
Change in cross-sectional area of the m. vastus lateralis of the quadriceps muscle | 8 weeks (+1-2 weeks) and 52 weeks (+1-2 weeks)
  By analysing muscle microbiopsies of the quadriceps muscle immunostaining of the myosin heavy chain, only for patients giving their specific consent.
Change in capillarisation of the m. vastus lateralis of the quadriceps muscle | 8 weeks (+1-2 weeks) and 52 weeks (+1-2 weeks)
  By analysing muscle microbiopsies of the quadriceps muscle, only for patients giving their specific consent.
Change in the amount of satellite cells of the m. vastus lateralis of the quadriceps muscle | 8 weeks (+1-2 weeks) and 52 weeks (+1-2 weeks)
  By analysing muscle microbiopsies with Pax7 immunostaining of the quadriceps muscle, only for patients giving their specific consent.
Change in gene expression of the m. vastus lateralis of the quadriceps muscle | 8 weeks (+1-2 weeks) and 52 weeks (+1-2 weeks)
  By analysing muscle microbiopsies with RT2 profiler PCR array skeletal muscle, Qiagen of the quadriceps muscle, only for patients giving their specific consent.
Minutes per day spent in at least moderate intense activities | 8 weeks and 52 weeks
  Change in minutes per day spent in at least moderate intense activities between baseline, 8 weeks and 52 weeks months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Mean walking time per day | 8 weeks and 52 weeks
  Change in mean daily walking time between baseline, 8 weeks and 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Mean sedentary time per day | 8 weeks and 52 weeks
  Change in mean sedentary time between baseline, 8 weeks and 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Daily number of steps at 8 weeks | 8 weeks
  Change in daily mean step count between baseline and 8 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Derom, Principal Investigator — UZ Gent; Wim Janssens, Principal Investigator — UZ Leuven; Heleen Demeyer, Principal Investigator — UGent; Thierry Troosters, Principal Investigator — KU Leuven; Marieke Wuyts, Principal Investigator — KU Leuven; Fien Hermans, Principal Investigator — U Gent
Locations (2):
- Belgium (2):
  - UZ Gent, Ghent
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data can be shared upon request.

REFERENCES:
- [Background] Wuyts M, Hermans F, Breuls S, Everaerts S, Derom E, Janssens W, Demeyer H, Troosters T. Development and feasibility of an exercise training program in primary care for patients with COPD experiencing an acute exacerbation. Physiotherapy. 2024 Jun;123:81-90. doi: 10.1016/j.physio.2023.09.003. Epub 2023 Oct 5. PMID 38295552